CLINICAL TRIAL: NCT03858205
Title: Phase II Multi-Institutional Study of Low-Dose (2Gy) Palliative Radiotherapy in the Treatment of Symptomatic Bone Metastases From Multiple Myeloma
Brief Title: Low-Dose Radiotherapy in Treating Painful Bone Metastases in Patients With Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16M-18-2; NCI-2018-03600 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16M-18-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2019-02-20; First posted 2019-02-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Bone Pain; Metastatic Malignant Neoplasm in the Bone; Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (low-dose radiation therapy) (Experimental): Patients receive low-dose radiation therapy at consecutive business days 1 and 2 in the absence of disease progression or unacceptable toxicity. Patients with no pain relief may receive additional radiotherapy at 4 weeks following initial radiotherapy.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Receive low-dose radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This phase II trial studies how well low-dose radiotherapy works in treating bone pain in patients with multiple myeloma that has spread to the bone. Radiation therapy uses high energy x-rays, gamma rays, neutrons, protons, or other sources to kill tumor cells and shrink tumors. Low-dose radiotherapy may be more convenient for patients and their families, may not interfere as much with the timing of chemotherapy, and may have less chance for short term or long-term side effects from the radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether treatment with 2 Gy x 2 to a painful myeloma bone lesion achieves patient-reported pain reduction comparable to current standard of care at 4 weeks.

SECONDARY OBJECTIVES:

I. To assess quality of life (QOL) in patients treated with 2 Gy x 2 to painful myeloma bone lesions.

II. To quantify analgesia use/reduction following 2 Gy x 2 to a painful myeloma bone lesion. All opioid analgesia use will be converted into morphine equivalent in order to compare across the entire population.

III. To measure time to pain relief and duration of pain relief with 2 Gy x 2.

EXPLORATORY OBJECTIVES:

I. To record cytogenetics and International Myeloma Working Group (IMWG) response criteria at diagnosis and prior to and following radiotherapy (RT).

OUTLINE:

Patients receive low-dose radiation therapy at consecutive business days 1 and 2 in the absence of disease progression or unacceptable toxicity. Patients with no pain relief may receive additional radiotherapy at 4 weeks following initial radiotherapy.

After completion of study treatment, patients are followed up at 2, 4, and 8 weeks and also at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of multiple myeloma
* Painful bone metastasis (index lesion) that has a radiographic correlate
* Patient may have had any number of prior chemotherapy/immunotherapy regimens (changes to systemic therapy or use of bisphosphonates for 4 weeks before and after RT are allowed, but recording of these changes must be made so it can be accounted for)
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Brief Pain Inventory (BPI) score >= 2
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients will be ineligible if the index lesion has received prior radiation therapy or prior palliative surgery. Patients may have received prior palliative or primary radiotherapy or surgery to other parts of the body, as long as the index lesion was not in the prior radiation fields and has not received prior palliative surgery
* Patients will also be ineligible if there is pathologic fracture or impending fracture at the site of the index lesion or planned surgical fixation of the bone at the index lesion
* Patients with clinical or radiographic evidence of spinal cord or cauda equina compression/effacement from the index lesion, and/or with index lesions located at the skull base or orbital lesions
* Patients must not be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2027-03-11 (Estimated)

PRIMARY OUTCOMES:
Pain response | Up to 6 months after completion of radiation therapy
  Pain will be measured using the Brief Pain Inventory (BPI).

SECONDARY OUTCOMES:
Quality of life (QOL) as measured by European Organization for Research and Treatment of Cancer Metastases Module (EORTC QLQ-BM22) | Up to 6 months after completion of radiation therapy
  Quality of life will be assessed before and after radiation therapy.
  EORTC QLQ-BM22 measures four multi-item scales: painful sites, functional interference, painful characteristics, and psychosocial aspects. Each item will be scaled as: 1= not at all; 2 = a little; 3 = quite a bit; 4 =very much. Answers will be converted into grading scale, with values between 0 and 100. Higher scores represent worse QOL for the subscales of painful sites, painful characteristics and psychosocial aspects, while higher scores in functional scale represents better functioning.
Quality of life (QOL) as measured by European Organization for Research and Treatment of Cancer Quality of life Questionnaire Core 30 (EORTC QLQ-C30) | Up to 6 months after completion of radiation therapy
  The QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item scales and single-item measures including functional scales, symptom scales, a global health status / QoL scale, and single item measures. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." The method for scoring these scales is: 1. Estimate the average of the items that contribute to the scale; this is the raw score. 2. Use a linear transformation to standardize the raw score, so that scores range from 0 to 100; a higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Garsa, MD, Principal Investigator — University of Southern California
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota - Masonic Cancer Center, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania